CLINICAL TRIAL: NCT04126681
Title: A Phase 2, Randomized, Open Label, Pivotal Study to Evaluate the Efficacy and Safety of HQP1351 in CML CP Patients Who Are Resistant and/or Intolerant to First- and Second-Generation Tyrosine Kinase Inhibitors
Brief Title: A Pivotal Study of HQP1351 in Patients With Chronic Myeloid Leukemia in Chronic Phase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: HealthQuest Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HQP1351CC203
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase
Keywords: Chronic Myeloid Leukemia; HQP1351; CML; CML-CP; Olverembatinib Tablets
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — olverembatinib; Hydroxyurea; Homoharringtonine; Imatinib Mesylate; Dasatinib; nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HQP1351 therapy cohort (Experimental): HQP1351 40 mg, taken orally once every other day of a 28-day cycle
  Interventions: Drug: HQP1351
- Best Available Therapy (BAT) cohort (Active Comparator): Best available therapy (BAT) will be selected by the investigator for each participant.
  Interventions: Drug: Hydroxyurea or Interferon-based therapy; Drug: Homoharringtonine; Drug: Imatinib, Dasatinib or Nilotinib

INTERVENTIONS:
Drug: HQP1351 — HQP1351 is a new, bioavailable inhibitor against BCRABLWT and a broad spectrum of BCR-ABL mutants including BCR-ABLT315I
  Arms: HQP1351 therapy cohort
Drug: Hydroxyurea or Interferon-based therapy — Patients will receive BAT based on the Investigator's opinion, taking into account the manufacturer's instructions, labeling, subject's medical condition, and institutional guidelines.
  Arms: Best Available Therapy (BAT) cohort
Drug: Homoharringtonine — Patients will receive BAT based on the Investigator's opinion, taking into account the manufacturer's instructions, labeling, subject's medical condition, and institutional guidelines.
  Arms: Best Available Therapy (BAT) cohort
Drug: Imatinib, Dasatinib or Nilotinib — Patients will receive BAT based on the Investigator's opinion, taking into account the manufacturer's instructions, labeling, subject's medical condition, and institutional guidelines.
  Arms: Best Available Therapy (BAT) cohort

SUMMARY:
The purpose of this study is to evaluate the efficacy of HQP1351 in patients with chronic myeloid leukemia in chronic phase (CML-CP) who are resistant and/or intolerant to first- and second-generation tyrosine kinase inhibitors. The efficacy of HQP1351 is determined by evaluating the subjects' event free survival (EFS).

DETAILED DESCRIPTION:
This is a phase 2, randomized, open label, pivotal study to evaluate the efficacy and safety of HQP1351 in CML CP patients who are resistant and/or intolerant to first- and second-generation TKIs in China. A total of 141 CML CP patients will be included in this study. After screening, eligible subjects will be randomized by 2:1 ratio to enter HQP1351 therapy cohort and best available therapy (BAT) cohort. When the subjects in the two cohorts reach EFS assessment, they can crossover to contralateral cohort if the investigator and Sponsor think they could be clinically benefited. During treatment, each subject will be assessed regularly for hematological, cytogenetic and molecular responses. At the same time, safety information also will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female patients who are 18 years of age or older.
2. CML-CP patients with positive Ph chromosome or BCR-ABL fusion genes.
3. Resistance and intolerance of first- and second-generation TKIs: defined as resistance or intolerance to imatinib, nilotinib, and dasatinib.
4. Ability to understand and willingness to sign a written informed consent form. The consent form must be signed by the patient prior to any study specific procedures.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
6. Predicted life expectancy of ≥3 months.
7. Organ function as indicated by the following laboratory indicators must be met (Hematological indicators require that no blood transfusion or any blood products or cytokines be used within 14 days prior to testing):

   * Hemoglobin ≥8.0g/dL.
   * White blood cell count ≥ 3.0×10^9/L.
   * Platelet count ≥ 75×10^9/L.
   * Serum creatinine ≤ 1.5×upper limit of normal (ULN) or 24 hours calculated creatinine clearance ≥ 50mL/min when serum creatinine >1.5×ULN.
   * Serum albumin ≥ 3.0 g/dL.
   * Total bilirubin ≤ 1.5 x ULN.
   * Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 x ULN.
   * Amylase≤1.5×ULN. Lipase≤1.5×ULN.
   * PT/APTT/INR≤1.5×ULN.
8. Cardiac function index: ejection fraction (EF) > 50%, pulmonary arterial systolic pressure (PASP) ≤50 mmHg.
9. QT interval corrected on electrocardiogram (ECG) evaluation: QTc≤450ms in males or ≤470ms in females.
10. Males and females of childbearing potential and their partners voluntarily take contraceptive measures that the researchers believe are effective within 120 days from the signing of the informed consent to the last use of the research drug, or confirm that sterilization has been performed (at least one month before screening).
11. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

1. Received cytotoxic chemotherapy or radiotherapy within 28 days prior to the first administration, interferon or cytarabine or antitumor effect Chinese herbal medicine or Chinese patent medicine within 14 days prior to the first administration, or targeted BCR-ABL1 TKI within 7 days prior to the first administration, or hydroxyurea or anagrelide within 24 hours after the first administration, or adverse events (except alopecia) caused by previous treatment and have not recovered.
2. The patients who received any other investigating drugs within 14 days prior to first administration.
3. For patients with CML-CP, if they have progressed to AP or BP, they cannot be enrolled after treatment with CML-CP.
4. Patients who are currently receiving treatment with a medication that has the potential to interact with research drug.
5. Have previously been treated with ponatinib or HQP1351 (or drugs of similar composition).
6. Absorption disorder syndrome or other diseases affecting oral drug absorption.
7. Have any history of heart or vascular disease, such as hypertension (systolic blood pressure (HBP) > 140mmHg and/or diastolic blood pressure > 90mmHg), or take medications that are known to cause QT interval prolongation. The patients with well controlled HBP can be included.
8. Pulmonary systolic pressure (PSP) of echocardiography is more than 50 mmHg, or there is clinical symptom related to pulmonary hypertension.
9. Have a history of serious cardiovascular diseases during the previous treatment of chronic myeloid leukemia with TKI, including myocardial infarction, unstable angina pectoris, severe arrhythmia and congestive heart failure.
10. Underwent autologous or allogeneic stem cell transplant.
11. CML-CP patient currently diagnosed as Complete cytogenetic response (CCyR).
12. Have diseases with abnormal bleeding and coagulation function, or have a bleeding disorder unrelated to CML within 3 months before first dose of study drug.
13. Underwent major surgery (except minor surgical procedures, such as placement or bone marrow biopsy) with 14 days prior to the first dose of study drug.
14. Require concurrent treatment with immunosuppressive agents, other than corticosteroids prescribed for a short course of therapy (It is defined as a daily dose of corticosteroids less than 30 mg prednisone or the same amount of other corticosteroids within 7 days).
15. Have active nervous system (CNS) disease as evidence by cytology or pathology. In the absence of clinical CNS disease, lumbar puncture is not required.
16. History of another primary malignancies.
17. Active symptomatic infection.
18. Known to be allergic to study drug ingredients or their analogues.
19. Female patients with blood β-Human chorionic gonadotropin positive, pregnant or lactating or expecting pregnancy during the study program.
20. Suffer from any condition or illness that, in the opinion of the Investigator or the medical monitor, would compromise patient safety or interfere with the evaluation of the safety of the research drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Event free survival (EFS) | By the end of Cycle 24 (each cycle is 28 days)
  EFS is defined as any "event" occurred since randomization, such as disease progression.

SECONDARY OUTCOMES:
Complete hematologic response (CHR) | By the end of Cycle 24 (each cycle is 28 days)
  CHR is the proportion of patients achieving CHR after being treated. It is defined as the best response obtained by the subjects during the whole treatment process of the study.
Major cytogenetic response (MCyR) | By the end of Cycle 24 (each cycle is 28 days)
  MCyR is the proportion of patients achieving Complete cytogenetic response (CCyR: defined as 0% Philadelphia chromosome-positive [Ph+] metaphases by cytogenetic analysis of bone marrow) or Partial Cytogenetic Response (PCyR: defined as >0% to 35% Ph+ metaphases by cytogenetic analysis of bone marrow). It is defined as the best response obtained by the subjects during the whole treatment process of the study.
Complete cytogenetic response (CCyR) | By the end of Cycle 24 (each cycle is 28 days)
  CCyR is the proportion of patients achieving CCyR after being treated. It is defined as the best response obtained by the subjects during the whole treatment process of the study.
Major molecular response (MMR) | By the end of Cycle 24 (each cycle is 28 days)
  MMR is the proportion of patients achieving a ratio of ≤0.1% breakpoint cluster region (BCR) abelson leukemia (ABL) to ABL transcripts on the international scale (≤0.1% BCR-ABL/ABL[IS]) after being treated with HQP1351. It is defined as the best response obtained by the subjects during the whole treatment process of the study.
Progression free survival (PFS) | By the end of Cycle 24 (each cycle is 28 days)
  PFS is defined as the interval between the first dose date and the first date at which the criteria for progression are met, or death. The subject who isn't progression or death will be censored at the last response assessment.
Overall survive (OS) | By the end of Cycle 24 (each cycle is 28 days)
  OS is defined as the interval between the first dose date and date of death, censored at the last contact date to be alive.
Incidence and severity of adverse events | By the end of Cycle 24 (each cycle is 28 days)
  Adverse events (AEs), and serious AEs (SAEs): Patients treatment related AE, SAE will be assessed according NCI CTCAE Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Huang, Professor, Principal Investigator — Peking University People's Hospital
Locations (22):
- China (22):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Gongdong
  - Nanfang hospital of southern medical university, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - The First affiliated hospital of Guangxi Medical University, Nanning, Guangxi
  - Henan Provincial Oncology Hospital, Zhengzhou, Henan
  - Henan Provincial people's Hospital, Zhengzhou, Henan
  - Tongji Hospital medical college Huazhong University of Science and Technology, Wuhan, Hubei
  - Union Hospital medical college Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First affiliated hospital of Nanchang University, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - The Affiliated hospital of Qingdao University, Qingdao, Shandong
  - Qilu hospital of Shandong University, Jinan, Shangdong
  - Ruijing Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine(hematology dept), Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine(HSCTdept), Hangzhou, Zhejiang

REFERENCES:
- [Derived] Jiang Q, Li Z, Qin Y, Li W, Xu N, Liu B, Zhang Y, Meng L, Zhu H, Du X, Chen S, Liang Y, Hu Y, Liu X, Song Y, Men L, Chen Z, Niu Q, Wang H, Lu M, Yang D, Zhai Y, Huang X. Olverembatinib (HQP1351), a well-tolerated and effective tyrosine kinase inhibitor for patients with T315I-mutated chronic myeloid leukemia: results of an open-label, multicenter phase 1/2 trial. J Hematol Oncol. 2022 Aug 18;15(1):113. doi: 10.1186/s13045-022-01334-z. PMID 35982483